CLINICAL TRIAL: NCT04209738
Title: Changes in Cardiovascular and Sleep Quality Parameters Under Eurythmy Therapy and Tai Chi in Comparison to Standard Care - a Substudy of the Multi-centre, Parallel-group, Randomised Controlled Trial to Assess the Efficacy and Safety of Eurythmy Therapy and Tai Chi in Comparison to Standard Care in Chronically Ill Elderly Patients With Increased Risk of Falling - ENTAiER Trial
Brief Title: Changes in Cardiovascular and Sleep Quality Parameters Under Eurythmy Therapy and Tai Chi in Comparison to Standard Care - A Substudy of the ENTAiER Trial
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EYT_12
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Fall Patients; Elderly Patients; Chronic Disease; Sleep Quality; Cardiovascular System; Tai Chi; Eurythmy Therapy
Keywords: Tai Chi; eurythmy; HRV; PWA; sleep quality; fall prevention
MeSH Terms: conditions — Chronic Disease; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eurythmy Therapy (performed as part of the ENTAiER main study): In group sessions á 5 patients with a qualified therapist: In the first 3 months 2 times a week, in the second 3 months once a week. Recommendation to practice at home at least 3 days a week (optimal to practice daily). They are supported by an eurythmy manual and an exercise video. This complements the regular care.
  Interventions: Other: This is an observational study being conducted as a substudy of another trial.
- Tai Chi (performed as part of the ENTAiER main study): In group sessions á 5 patients with a qualified teacher: In the first 3 months 2 times a week, in the second 3 months once a week. Recommendation to practice at home at least 3 days a week (optimal to practice daily). They are supported by a Tai Chi manual and a practice video. This complements the regular care.
  Interventions: Other: This is an observational study being conducted as a substudy of another trial.
- Standard Care: Brochure with detailed description of different evidence-based measures for fall prevention, created for the specific age group ("Gleichgewicht & Kraft - Trittsicher durchs Leben "https://www.trittsicher.org/files/trittsicher_bzga_sturzpraevention_2015-11-23.pdf") and recommendation to visit the family doctor and discuss fall prophylaxis with him.
  Interventions: Other: This is an observational study being conducted as a substudy of another trial.

INTERVENTIONS:
Other: This is an observational study being conducted as a substudy of another trial. — This is an observational study being conducted as a substudy of another trial. No intervention is planned for Substudy.

SUMMARY:
ENTAiER study is a multicentre randomized controlled trial to assess the efficacy and safety of eurythmy therapy and Tai Chi in comparison to standard care in chronically ill elderly patients with increased risk of falling. Subjects will be randomized to eurythmy therapy or Tai Chi or standard care alone. To investigate the changes in cardiovascular and sleep quality parameters under Eurythmy Therapy and Tai Chi in comparison to Standard Care in this trial, a substudy will be conducted only at the ARCIM Institute. The substudy will recruit enrolled participants from the ENTAiER trial to record various cardiovascular and sleep quality parameters. The aim is to compare changes in cardiovascular and sleep quality parameters under eurythmy therapy, Tai Chi and standard care alone in chronically ill elderly patients with increased risk of falling.

DETAILED DESCRIPTION:
This is an optional substudy of a multi-centre, parallel-group, three-arm randomized controlled trial - ENTAiER trial - to compare the changes in cardiovascular and sleep quality parameters under Eurythmy Therapy and Tai Chi in comparison to Standard Care in chronically ill elderly patients with increased risk of falling (see DRKS-ID: DRKS00016609). Subjects who consent to enroll in ENTAiER will be asked to participate in this substudy. The main focus of this substudy is on assessing the effects of Tai Chi and Eurythmy on the vegetative nervous system by measuring various parameters of heart rate variability and pulse wave analysis. In addition, the effects on sleep quality will be assessed. Participants of the substudy will undergo a measurement of heart rate variability with a long-term-ECG (Bittium Faros 360 TM), a pulse wave analysis, recorded with a vital function monitor (VitaGuard® 3100 monitor, getemed, Germany), and a blood pressure measurement and they fill in a sleep quality questionnaire (Pittsburgh Sleep Quality Index, PSQI) at baseline and after 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this substudy, subjects must be enrolled in ENTAiER main study and provide separate written informed consent for EYT_12 Substudy. See DRKS-ID: DRKS00016609 for inclusion criteria into ENTAiER main study

Exclusion Criteria for Substudy:

* Cardiac pacemaker
* Atrial fibrillation (documented in medical reports)
* To be eligible for this substudy, subjects must be enrolled in ENTAiER main study and provide separate written informed consent for EYT_12 Substudy. See DRKS-ID: DRKS00016609 for exclusion criteria into ENTAiER main study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects who have consented to participate and are enrolled in ENTAiER main study will be approached for participation in this substudy. Substudy will be conducted at the ARCIM Institute, Filderstadt.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Change in RMSSD | Continuous measurement (up to 15 minutes) at Baseline (pre-intervention) and 6 month (post-intervention)
  Root Mean Square of Successive Differences (ms), assessed with 24h ECG recorder Bittium Faros 360™, continuous measurement (up to 15 minutes) during standardized rest period at Baseline (pre-intervention) and 6 month (post-intervention)

SECONDARY OUTCOMES:
HRV analysis: Change in SDNN | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Standard deviation of normal to normal (NN) intervals (ms), assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in pNN50 | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Percentage of successive NN intervals that differ from each other by more than 50 ms (%), assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in HF | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  High frequency power band (0.15-0.40 Hz) (ms2) from frequency domain analysis, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in LF | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Low frequency power band (0.04-0.15 Hz) (ms2) from frequency domain analysis, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in LF/HF ratio | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  LF/HF ratio = ratio of the power in the LF band to the power in the HF band, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in VLF | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Very low frequency power band (0.00-0.04 Hz) (ms2) from frequency domain analysis , assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in MEAN HR [1/MIN] | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Mean Heart Rate, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
Change in HRV analysis: Change in SD2/SD1 RATIO | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Ratio of SD2 (standard deviation in long term of the RR interval) to SD1 (standard deviation of instantaneous beat-by beat variability), assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in STRESSINDEX | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Stress index (SI), assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in RESP. RATE | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Respiratory rate, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in HEART RATE / RESP. RATE RATIO | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Ratio of Heart Rate to Respiratory rate, assessed with 24h ECG Bittium Faros 360 TM, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
Pulse wave analysis: Change in Stiffness Index | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Stiffness Index, assessed with VitaGuard® 3100 monitor, getemed, Germany, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
Pulse wave analysis: Change in Reflection Index | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Reflection Index (RI, %), assessed with VitaGuard® 3100 monitor, getemed, Germany, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
Pulse wave analysis: Change in Perfusion Index | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Perfusion Index (PI, %), assessed with VitaGuard® 3100 monitor, getemed, Germany, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
Pulse wave analysis: Change in Pulse Transit Time | Continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Pulse Transit Time (PTT-W1, ms), assessed with VitaGuard® 3100 monitor, getemed, Germany, continuous measurement (up to 15 minutes) during standardized rest period at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
HRV analysis: Change in RMSSD | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Root Mean Square of Successive Differences (ms), assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in SDNN | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Standard deviation of normal to normal (NN) intervals (ms), assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in pNN50 | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Percentage of successive NN intervals that differ from each other by more than 50 ms (%), assessed with 24h ECG recorder Bittium Faros 360™ continuous 24-hour measurement measured for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in HF | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  High frequency power band (0.15-0.40 Hz) (ms2) from frequency domain analysis, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement measured for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in LF | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Low frequency power band (0.04-0.15 Hz) (ms2) from frequency domain analysis, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in LF/HF ratio | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  LF/HF ratio = ratio of the power in the LF band to the power in the HF band, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in VLF | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Very low frequency power band (0.00-0.04 Hz) (ms2) from frequency domain analysis, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in MEAN HR [1/MIN] | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Mean Heart Rate, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in SD2/SD1 RATIO | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Ratio of SD2 (standard deviation in long term of the RR interval) to SD1 (standard deviation of instantaneous beat-by beat variability), assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in STRESSINDEX | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Stress index (SI), assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
Change in HRV analysis: RESP. RATE | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Respiratory rate, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
HRV analysis: Change in HEART RATE / RESP. RATE RATIO | Continuous 24-hours measurement at baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Ratio of Heart Rate to Respiratory rate, assessed with 24h ECG recorder Bittium Faros 360™, continuous 24-hour measurement for day and night phase at Baseline (pre-intervention) and 6 month (post-intervention)
Change in SBP | Baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Systolic Blood Pressure
Change in DBP | Baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Diastolic Blood Pressure
24h activity protocol: change in sleep quality | Baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Self-reported sleep quality during the night after application of the long-term ECG, assessed with a 10-point scale (1=bad, 10=good)
Change in PSQI | Baseline (t0), 3 month (t1), 6 month (t2) and 12 month (t3)
  Pittsburgh Sleep Quality Index (PSQI): Total Score. The PSQI is a validated self-rating instrument assessing aspects of sleep quality.Minimum score 0 (better); maximum score 21 (worse) < or = 5 associated with good sleep quality; > 5 associated with poor sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Study Director — ARCIM Institute Academic Research in Complementary and Integrative Medicine
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.